CLINICAL TRIAL: NCT01543308
Title: Phase 1 Study of Coronary Heart Disease Proteomics Research
Brief Title: The Alteration of HDL Protein Composition in Patients With Coronary Heart Disease Before and After Statins Treatment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government); Beijing Proteome Research Center (Other)
Responsible Party: Principal Investigator, Yan Li-rong, Key Laboratory of Clinical Trial Research in Cardiovascular Drugs, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2011-HDL-01
Record Dates: First submitted 2012-02-21; First posted 2012-03-02 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — frozen in -80C
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- coronary heart disease
- healthy control group

SUMMARY:
The protein composition of HDL is complicated. The investigators have identified 40 distinct proteins associated with HDL by proteomics technology, and these proteins have been confirmed to be related to the function of anti-inflammation, anti-oxidation, improvement of endothelial function, inhibition of thrombosis and so on. And the investigators also found that the levels of some proteins in HDL changed in patients with coronary heart disease, compared with the healthy control group.

So, this study is to conduct in the two following aspects: enlarge the sample size to verify the preliminary results to find new research ideas of pathogenesis and biomarkers for coronary heart disease; and study the changes of HDL protein composition in patients with coronary heart disease before and after statins treatment using proteomics technology in order to find the mechanism of statins pleiotropic effects and indicators for evaluating the treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

Angiographic evidence of coronary artery disease, and no lipid-lowering therapy in the past 2 weeks for treatment group;

Exclusion Criteria:

* Use of potent lipid-lowering therapy for more than 2 weeks; myocardial infarction or percutaneous coronary intervention in the past 6 months; severe congestive heart failure, valvular heart disease and other non-coronary heart disease cardiovascular disease; liver or renal dysfunction; connective tissue disease; infection, Malignancy; and other conditions that physicians considered inappropriate to the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinical indication for coronary heart disease and no lipid-lowering therapy in the past 2 weeks
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Differential Proteins and the levels of Differential Proteins | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hong Liu, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Key Laboratory of Clinical Trial Research in Cardiovascular Drugs, FuWai Hospital, Beijing, China